CLINICAL TRIAL: NCT00973154
Title: Corticosteroid Treatment for Community-Acquired Pneumonia A Randomized, Double-blind Study- The STEP Trial
Brief Title: Corticosteroid Treatment for Community-Acquired Pneumonia - The STEP Trial
Acronym: STEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Kantonsspital Aarau (Other); Kantonsspital Liestal (Other)
Responsible Party: Principal Investigator, Mirjam Christ-Crain, Prof. Dr. med. Leitende Aerztin, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STEP
Record Dates: First submitted 2009-09-07; First posted 2009-09-09 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2014-05

CONDITIONS: Community-acquired Pneumonia
Keywords: Pneumonia; Corticosteroids; clinical stability
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Active Comparator): Drug
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — 50mg per day of prednisone orally for 7 days versus placebo

SUMMARY:
Background: An intact hypothalami-pituitary-adrenal (HPA) axis with an effective intracellular anti-inflammatory activity of glucocorticoids is indispensable for host survival during stress upon exposure to an infectious agent. Community-acquired pneumonia (CAP) is characterized by significant mortality and increased circulating inflammatory cytokines. Despite adequate antimicrobial therapy mortality rates for CAP have not changed over several decades. The use of corticosteroids in patients with CAP is inconclusive.

Study aim: To compare a 7 days treatment with prednisone and placebo in patients with community-acquired pneumonia with respect to time to clinical stability.

Study hypothesis: The investigators hypothesize that use of corticosteroids will lead to a 25% relative risk reduction for death and clinical instability.

Study type: randomized double blind intervention study

Patients: 800 patients with community-acquired pneumonia

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older admitted for hospitalization from the community or a nursing home with CAP.
2. CAP will be defined by a new infiltrate on chest radiograph and the presence of one or several of the following acute respiratory signs or symptoms:

   * cough
   * sputum production
   * dyspnea
   * core body temperature >38.0° C
   * auscultatory findings of abnormal breath sounds and rales
   * leukocyte count >10 or <4 x 109 cells L-1 (1)

Exclusion Criteria:

1. Patients or family members unable to give written informed consent, e.g. with severe dementia.
2. Patients with active intravenous drug use.
3. Severe immunosuppression (e.g. patients infected with human immunodeficiency virus infection and a CD4 count below 350 x 109/L, patients on immunosuppressive therapy after solid organ transplantation and neutropenic patients with neutrophil count < 500 x 109/L and patients under chemotherapy with neutrophils 500-1000 x 109/L with an expected decrease to values < 500 x 109/L); patients with cystic fibrosis as well as patients with active tuberculosis.
4. Patients with acute burn injury
5. Patients with acute gastrointestinal bleeding within 3 months of the current hospitalization
6. Patients with an acute concomitant condition requiring more than 0.5mg/kg/d prednisone equivalent
7. Pregnancy or breast feeding
8. Patients with known adrenal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2009-12; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time to clinical stability | 30 days

SECONDARY OUTCOMES:
Side effects of corticosteroids, mortality, recurrence | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (7):
- Switzerland (7):
  - Medizinische Klinik, Kantonsspital Liestal, Liestal, Basel-Landschaft
  - Medicine Interne, Hôpital du Jura, site de Delémont, Delémont, Canton of Jura
  - Kantonsspital Aarau, Aarau
  - University Hospital Basel, Basel
  - Inselspital, Bern
  - Bruderholzspital, Bruderholz
  - Bürgerspital, Solothurn

REFERENCES:
- [Derived] Blum CA, Roethlisberger EA, Cesana-Nigro N, Winzeler B, Rodondi N, Blum MR, Briel M, Mueller B, Christ-Crain M, Schuetz P. Adjunct prednisone in community-acquired pneumonia: 180-day outcome of a multicentre, double-blind, randomized, placebo-controlled trial. BMC Pulm Med. 2023 Dec 11;23(1):500. doi: 10.1186/s12890-023-02794-w. PMID 38082273
- [Derived] Borisov AN, Blum CA, Christ-Crain M, Ebrahimi F. No obesity paradox in patients with community-acquired pneumonia - secondary analysis of a randomized controlled trial. Nutr Diabetes. 2022 Mar 23;12(1):12. doi: 10.1038/s41387-022-00190-7. PMID 35322019
- [Derived] Sailer CO, Refardt J, Blum CA, Schnyder I, Molina-Tijeras JA, Fenske W, Christ-Crain M. Validity of different copeptin assays in the differential diagnosis of the polyuria-polydipsia syndrome. Sci Rep. 2021 May 12;11(1):10104. doi: 10.1038/s41598-021-89505-9. PMID 33980941
- [Derived] Potasso L, Sailer CO, Blum CA, Cesana-Nigro N, Schuetz P, Mueller B, Christ-Crain M. Mild to moderate hyponatremia at discharge is associated with increased risk of recurrence in patients with community-acquired pneumonia. Eur J Intern Med. 2020 May;75:44-49. doi: 10.1016/j.ejim.2019.12.009. Epub 2020 Jan 15. PMID 31952985
- [Derived] Popovic M, Cesana-Nigro N, Winzeler B, Thomann R, Schutz P, Muller B, Christ-Crain M, Blum CA. Estimation of treatment allocation in a randomised, double-blinded, placebo-controlled trial. Swiss Med Wkly. 2019 Jul 24;149:w20114. doi: 10.4414/smw.2019.20114. eCollection 2019 Jul 15. PMID 31340056
- [Derived] Blum CA, Schuetz P, Nigro N, Winzeler B, Arici B, Refardt J, Urwyler SA, Rodondi N, Blum MR, Briel M, Mueller B, Christ-Crain M. Cosyntropin testing does not predict response to glucocorticoids in community-acquired pneumonia in a randomized controlled trial. Clin Endocrinol (Oxf). 2019 Sep;91(3):374-382. doi: 10.1111/cen.13907. Epub 2019 Jan 9. PMID 30485501
- [Derived] Popovic M, Blum CA, Nigro N, Mueller B, Schuetz P, Christ-Crain M. Benefit of adjunct corticosteroids for community-acquired pneumonia in diabetic patients. Diabetologia. 2016 Dec;59(12):2552-2560. doi: 10.1007/s00125-016-4091-4. Epub 2016 Sep 10. PMID 27614658
- [Derived] Wirz SA, Blum CA, Schuetz P, Albrich WC, Noppen C, Mueller B, Christ-Crain M, Tarr PE; STEP Study Group. Pathogen- and antibiotic-specific effects of prednisone in community-acquired pneumonia. Eur Respir J. 2016 Oct;48(4):1150-1159. doi: 10.1183/13993003.00474-2016. Epub 2016 Jul 28. PMID 27471201
- [Derived] Blum CA, Nigro N, Briel M, Schuetz P, Ullmer E, Suter-Widmer I, Winzeler B, Bingisser R, Elsaesser H, Drozdov D, Arici B, Urwyler SA, Refardt J, Tarr P, Wirz S, Thomann R, Baumgartner C, Duplain H, Burki D, Zimmerli W, Rodondi N, Mueller B, Christ-Crain M. Adjunct prednisone therapy for patients with community-acquired pneumonia: a multicentre, double-blind, randomised, placebo-controlled trial. Lancet. 2015 Apr 18;385(9977):1511-8. doi: 10.1016/S0140-6736(14)62447-8. Epub 2015 Jan 19. PMID 25608756
- [Derived] Blum CA, Nigro N, Winzeler B, Suter-Widmer I, Schuetz P, Briel M, Bingisser R, Zimmerli W, Ullmer E, Elsaesser H, Tarr P, Wirz S, Thomann R, Hofmann E, Rodondi N, Duplain H, Burki D, Mueller B, Christ-Crain M. Corticosteroid treatment for community-acquired pneumonia--the STEP trial: study protocol for a randomized controlled trial. Trials. 2014 Jun 28;15:257. doi: 10.1186/1745-6215-15-257. PMID 24974155